CLINICAL TRIAL: NCT06536309
Title: Neprilysin Inhibition to Reduce Myocardial Fibrosis in Heart Failure With Preserved Ejection Fraction
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Jonathan Cunningham MD MPH, Assistant Professor of Medicine, Cardiovascular Division, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2024P001894; 1K23HL168163-01A1 (NIH)
Record Dates: First submitted 2024-07-26; First posted 2024-08-02 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Heart Failure With Preserved Ejection Fraction; Myocardial Fibrosis
MeSH Terms: interventions — sacubitril and valsartan sodium hydrate drug combination; Valsartan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Sacubitril/valsartan (Experimental): Patient randomized to the interventional arm will be treated with sacubitril/valsartan
  Interventions: Drug: Sacubitril-valsartan
- Valsartan (Active Comparator): Patient randomized to the active comparator arm will be treated with valsartan
  Interventions: Drug: Valsartan

INTERVENTIONS:
Drug: Sacubitril-valsartan — Sacubitril-valsartan titrated to maximally targeted dose
  Other Names: Entresto
  Arms: Sacubitril/valsartan
Drug: Valsartan — Valsartan titrated to maximally targeted dose
  Other Names: Diovan
  Arms: Valsartan

SUMMARY:
Cardiac magnetic resonance imaging (MRI) measures of myocardial interstitial fibrosis (MIF) are elevated in heart failure with preserved ejection fraction (HFpEF) patients and associated with poor prognosis. Extracellular volume (ECV) is the most reproducible and best validated cardiac MRI measure of MIF. Sacubitril/valsartan reduces histological MIF in mice and levels of some extracellular matrix regulatory proteins in humans with HFpEF. However, the effect of sacubitril/valsartan on robust measures of MIF in humans is unknown. Demonstrating reductions in ECV with sacubitril/valsartan would clarify the mechanism of this approved medication. Given the borderline reduction in heart failure hospitalizations with sacubitril/valsartan and the heterogeneity of HFpEF pathophysiology, this result would suggest that neprilysin inhibition may particularly benefit HFpEF patients with greater MIF. The investigators propose a proof-of-concept clinical trial to evaluate the effect of neprilysin inhibition (sacubitril/valsartan vs valsartan alone) on cardiac MRI measures of fibrosis (principally ECV) and circulating protein levels.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 50 years or older
* Able to provide informed consent, as assessed by a physician investigator, and willing to comply with the study
* Clinically confirmed diagnosis of heart failure
* Left ventricular ejection fraction greater than or equal to 45% within 1 year by echocardiogram, cardiac MRI, or nuclear scan

Exclusion Criteria:

* Contraindication to MRI (metal prosthesis, implantable cardiac device, or severe claustrophobia)
* Systolic blood pressure < 100mm Hg, or <110 mm Hg for patients not taking an ACE inhibitor or angiotensin receptor blocker
* symptomatic hypotension
* eGFR < 30 mL/min/1.73m2 within 60 days of enrollment
* Serum potassium >5.2mmol/L within 60 days of enrollment, or >5.0 mmol/L for patients not taking an ACE inhibitor or angiotensin receptor blocker
* Myocardial infarction within 6 months of enrollment
* Infiltrative or hypertrophic cardiomyopathy
* History of cirrhosis, biliary cirrhosis, or cholestasis
* History of angioedema
* Pregnancy, planning pregnancy, or breastfeeding
* Active treatment with lithium or a direct renin inhibitor

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
Change in extracellular volume by cardiac MRI | 1 year
  The primary outcome is to evaluate the change in extracellular volume (ECV), measured by cardiac MRI, from baseline to one year, in the sacubitril/valsartan arm compared to the valsartan arm

SECONDARY OUTCOMES:
Change in left ventricular native T1 time | 1 year
  Measured by cardiac MRI

OTHER OUTCOMES:
Change in left ventricular mass | 1 year
  Measured by cardiac MRI
Change in left atrial size | 1 year

IPD SHARING:
Plan to Share IPD: No
Deidentified participant data will be made available according to NHLBI and institutional regulations

REFERENCES:
- [Background] Solomon SD, McMurray JJV, Anand IS, Ge J, Lam CSP, Maggioni AP, Martinez F, Packer M, Pfeffer MA, Pieske B, Redfield MM, Rouleau JL, van Veldhuisen DJ, Zannad F, Zile MR, Desai AS, Claggett B, Jhund PS, Boytsov SA, Comin-Colet J, Cleland J, Dungen HD, Goncalvesova E, Katova T, Kerr Saraiva JF, Lelonek M, Merkely B, Senni M, Shah SJ, Zhou J, Rizkala AR, Gong J, Shi VC, Lefkowitz MP; PARAGON-HF Investigators and Committees. Angiotensin-Neprilysin Inhibition in Heart Failure with Preserved Ejection Fraction. N Engl J Med. 2019 Oct 24;381(17):1609-1620. doi: 10.1056/NEJMoa1908655. Epub 2019 Sep 1. PMID 31475794